CLINICAL TRIAL: NCT01010438
Title: Clinical Evaluation of an Apnea Index Provided by a Capnograph/Pulse Oximeter to Assist in the Diagnosis and Screening of Obstructive Sleep Apnea
Brief Title: Clinical Evaluation of an Apnea Index for Diagnosis and Screening of Obstructive Sleep Apnea (OSA)
Status: Completed | Type: Observational
Sponsor: Oridion (Industry)
Responsible Party: Sponsor
Organization: Medtronic - MITG (Industry)
Other Study IDs: D006567
Record Dates: First submitted 2009-11-08; First posted 2009-11-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep studies; sleep apnea; OSA; Referred for sleep studies by a medical professional
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adults: Adult patients referred for sleep studies, including both patients with suspected OSA and patients that have been invited to a sleep lab for reasons not related to OSA such as insomnia, para-insomnia and similar.
- Children (1-17): Pediatric patients referred for sleep studies, including both patients with suspected OSA and patients that have been invited to a sleep lab for reasons not related to OSA such as insomnia, para-insomnia and similar.

SUMMARY:
The study is designed to compare the apnea event recognition capability of the Capnostream 20 with investigational software to polysomnograph recordings scored by a trained analyst. The study will compare the apnea index score (AI) calculated by the Capnostream 20 algorithm based on capnography to that calculated by a trained analyst evaluating polysomnograph recordings.

To this aim, subjects will be connected to EMBLA N7000 Polysomnograph, and to the Capnostream 20, in order to monitor CO2 and SpO2 during routine overnight sleep studies.

The Capnostream, using both its USB Data Port and Analog output port will simultaneously provide the monitored data both to a USB flash memory device and Polysomnograph for storage for future analysis.

The data collected by the Polysomnograph including the Capnostream data will be analyzed by a trained expert for evaluation of apnea events obtained from both sources.

In parallel, the Capnostream data as collected with the USB flash memory, will be downloaded onto a PC, and using the Oridion software algorithm designed for evaluating the data (to be implemented in the monitor when validated), the Apnea Index and Oxygen Desaturation Index will be calculated. The results of the Apnea Index scores calculated from the Polysomnograph and from the DUT will be compared.

Based on the results, the study will then evaluate the ability of the Capnograph/Pulse-Oximeter as a tool for screening and assisting in the diagnosis of patients with obstructive sleep-apnea in the hospital environment, where it is being used as a ventilation monitor based on the demonstration of a high correlation with the gold standard in the sleep lab.

DETAILED DESCRIPTION:
The clinical investigation will be conducted until enrollment of at least 30 adult and 30 Pediatric patients of both sexes with complete data sets are collected from three different sleep lab sites per the FDA guidance requirements. The enrollment time will last up to six (6) months. The overall number of enrolled patients (i.e. with complete/incomplete data) will not exceed 80 patients.

ELIGIBILITY:
Inclusion Criteria:

* All Adults > 18 years old and able to understand and give consent per the IRB or a child above one years old consented by a parent or legal guardians.
* Patients consented or for whom legal guardians consented for the participation of this trial.
* Patient recommended for a Sleep assessment by medical staff.

Exclusion Criteria:

* Patients who in the opinion of the investigator should not participate.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population includes consented adult patients and pediatric patients from 3 sites that have been referred for sleep studies by a medical professional. The study will include both patients with suspected OSA and patients that have been invited to a sleep lab for reasons not related to OSA such as insomnia, para-insomnia and similar.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Comparison of apnea event detection | Apnea events are defined as events that last at least 10 seconds

SECONDARY OUTCOMES:
Validation of apnea index | Post study analysis

CONTACTS AND LOCATIONS:
Overall Officials: Giora Pillar, MD, Principal Investigator — Deputy Director, Department of Pediatrics, Director, Pediatric Sleep Disorders Unit, Rambam Health Care Campus
Locations (3):
- Israel (3):
  - Hillel Yaffe Sleep Lab Center, Hadera
  - Prof. Giora Pillar M.D., Deputy Director, Department of Pediatrics, Director, Pediatric Sleep Disorders Unit, Haifa
  - Hadassah Sleep Lab Center, Jerusalem

REFERENCES:
- [Background] Dangers of Postoperative Opioids - APSF Workshop and White Paper Address Prevention of Postoperative Respiratory Complications /Matthew B. Weinger, MD/APSF Newsletter Volume 21, No. 4, 61-88Winter 2006-2007
- [Background] The AASM Manual for the Scoring of Sleep and Associated Events: Rules, Terminology and Technical Specification/ Con Iber, MD/ AASM - 2007
- [Background] Ng SS, Chan TO, To KW, Ngai J, Tung A, Ko FW, Hui DS. Validation of a portable recording device (ApneaLink) for identifying patients with suspected obstructive sleep apnoea syndrome. Intern Med J. 2009 Nov;39(11):757-62. doi: 10.1111/j.1445-5994.2008.01827.x. Epub 2008 Nov 3. PMID 19220528
- [Background] de Almeida FR, Ayas NT, Otsuka R, Ueda H, Hamilton P, Ryan FC, Lowe AA. Nasal pressure recordings to detect obstructive sleep apnea. Sleep Breath. 2006 Jun;10(2):62-9. doi: 10.1007/s11325-005-0042-x. PMID 16502297